CLINICAL TRIAL: NCT06996665
Title: Diaphragmatic Physiology Similarity Index May Titrate HFNC Flow Setting: A Prospective Observational Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Huiqing Ge, Director of Respiratory Medicine, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20250271
Record Dates: First submitted 2025-05-03; First posted 2025-05-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Failure
Keywords: Diaphragm; Speckle Tracking; PEEP
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Feasibility Patient Cohort（No Intervention / Diagnostic Test） (No Intervention): Participants undergo an assessment-only diagnostic intervention: diaphragmatic speckle-tracking ultrasound performed at predefined time points during routine care to evaluate feasibility and measurement properties (e.g., foundational speckle-tracking metrics and inter-/intra-operator reproducibility). Images of the bilateral zone of apposition are acquired and analyzed offline for the contraction synchrony index, end-diaphragmatic residual contraction (EDRC), displacement velocity, and maximal displacement. Ultrasound findings are not used for clinical decision-making; respiratory support (e.g., HFNC/ventilator settings) is determined independently by the treating clinicians.
- Healthy Volunteer Reference Cohort (No Intervention): Healthy volunteers undergo protocolized, assessment-only diaphragmatic speckle-tracking ultrasound to characterize normal diaphragmatic physiology and establish reference ranges; no feasibility or reproducibility endpoints are collected. Bilateral zone-of-apposition images are acquired and analyzed offline for DPSI, contraction synchrony index, end-diaphragmatic residual contraction (EDRC), displacement velocity, and maximal displacement. No therapeutic interventions are delivered, and participation does not alter clinical management.
- Sequence 1: 20-30-40-60 L/min (Experimental): Participants receive HFNC flows 20→30→40→60 L/min across four periods. Each period maintains the assigned flow for a predefined steady window; FiO₂ is adjusted per routine to meet target SpO₂. At the end of each period, protocolized diaphragmatic speckle-tracking ultrasound (bilateral zone of apposition) is performed with offline analysis of DPSI, contraction synchrony index, EDRC, displacement velocity, and maximal displacement; vital signs, respiratory rate, comfort/tolerance, and oxygenation are recorded. Safety overrides (e.g., hypoxemia, distress, intolerance) permit clinicians to modify or terminate the period.
  Interventions: Other: High-flow adjustment sequence
- Sequence 2: 30-60-20-40 L/min (Experimental): This sequence administers HFNC flows 30→60→20→40 L/min over four periods. Procedures mirror Sequence 1: predefined steady windows, routine FiO₂ titration, end-of-period speckle-tracking ultrasound with offline metrics (DPSI, synchrony, EDRC, displacement velocity, maximal displacement), and collection of vitals/oxygenation/tolerance; safety triggers allow clinical override.
  Interventions: Other: High-flow adjustment sequence
- Sequence 3: 40-20-60-30 L/min (Experimental): Participants receive HFNC flows 40→20→60→30 L/min across four periods. A predefined steady window is maintained with routine FiO₂ adjustments. End-of-period speckle-tracking ultrasound is performed with the same offline metrics; vitals, respiratory rate, comfort/tolerance, and oxygenation are captured. Safety triggers enable clinical override.
  Interventions: Other: High-flow adjustment sequence
- Sequence 4: 60-40-30-20 L/min (Experimental): HFNC flows are delivered 60→40→30→20 L/min over four periods. Each period preserves a steady observation window with routine FiO₂ titration; end-of-period speckle-tracking ultrasound is performed with offline analyses (DPSI, synchrony, EDRC, displacement velocity, maximal displacement), and vitals/oxygenation/tolerance are recorded. Safety overrides may be applied by the treating team.
  Interventions: Other: High-flow adjustment sequence

INTERVENTIONS:
Other: High-flow adjustment sequence — Delivers heated, humidified blended oxygen via HFNC with real-time titration based on diaphragmatic speckle-tracking metrics (e.g., DPSI, contraction synchrony). Flow is adjusted in predefined increments to reach target diaphragmatic physiology while FiO₂ is titrated to maintain target SpO₂. Ultrasound feedback is used for bedside decisions; safety triggers allow clinical override.
  Arms: Sequence 1: 20-30-40-60 L/min; Sequence 2: 30-60-20-40 L/min; Sequence 3: 40-20-60-30 L/min; Sequence 4: 60-40-30-20 L/min

SUMMARY:
Study Objective This prospective observational study aims to investigate the role of the Diaphragmatic Physiology Similarity Index (DPSI) derived from speckle tracking ultrasound in titrating high-flow nasal cannula (HFNC) flow settings, and to evaluate its application in patients with acute respiratory failure.

Primary Research Questions

To characterize the features of the DPSI in healthy individuals and in patients with acute respiratory failure.

To assess the behavior of the DPSI under different HFNC flow settings in patients with acute respiratory failure.

Secondary Research Questions

Feasibility and inter-operator reproducibility of diaphragmatic speckle tracking.

Assessment of the Diaphragmatic Contraction Synchrony Index.

Evaluation of End-Diaphragmatic Residual Contraction (EDRC).

Additional fundamental parameters, including diaphragmatic displacement velocity and maximum displacement.

ELIGIBILITY:
Feasibility and reproducibility：adult ICU patients

Methodology for diaphragmatic motion synchrony:healthy adults and adult ICU patients Between-group comparisons and flow-titration study

Inclusion Criteria:

1. Age ≥18 years old.
2. Clear diagnosis of respiratory failure requiring respiratory support.
3. Expected duration of respiratory support ≥24 hours or (high-flow/non-invasive ventilation) ≥48 hours.
4. Voluntary participation in this study and signed informed consent. If the participant is unable to read or sign the informed consent form due to incapacity (e.g., unconsciousness), the legal guardian must act as a proxy in the informed consent process and sign the form. If the participant cannot read the consent form (e.g., illiterate participants), a witness must observe the informed consent process and sign the form.

Exclusion Criteria:

1. Severe chest wall deformities or diaphragmatic paralysis.
2. End-stage disease with a predicted life expectancy of less than 24 hours.
3. Inability to acquire STE (strains and echoes) images (e.g., severe subcutaneous emphysema, position limitations).
4. Vulnerable groups other than critically ill patients/elderly/illiterate individuals, including those with mental disorders, cognitive impairments, pregnant women, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic Physiology Similarity Index (DPSI) | Healthy Participants: Baseline； Baseline evaluation at the time of enrollment change with each change in ventilation parameters.
  The objective of this prospective observational study is to explore the Diaphragmatic Physiology Similarity Index (DPSI), derived from speckle tracking ultrasound, in guiding the adjustment of high-flow nasal cannula (HFNC) flow settings, and to assess its application in patients with acute respiratory failure.

SECONDARY OUTCOMES:
Adverse events including pneumothorax, hemodynamic instability, and other complications | At baseline (upon enrollment), 1 hour / 6 hours / 24 hours after intervention, and during daily morning assessments until extubation or day 28.
Arterial blood gas analysis (ABG analysis) | At baseline (upon enrollment), 1 hour / 6 hours / 24 hours after intervention, and during daily morning assessments until extubation or day 28.
Diaphragmatic Contraction Synchrony Index | After each HFNC flow adjustment: Measure contraction synchrony during each flow setting period.
  Evaluate the diaphragmatic contraction synchrony index, assessing the degree to which the diaphragm contracts as a coordinated unit.
ICC (Intraclass Correlation Coefficient) | At each ultrasound assessment, record the percentage of analyzable images. Compare measurements at the beginning and throughout the study among operators.
  Evaluate the feasibility and inter-operator reproducibility of diaphragmatic speckle tracking ultrasound.
Evaluation of End-Diaphragmatic Residual Contraction (EDRC) | After each mechanical ventilation period: Measure EDRC at the end of the mechanical ventilation phase, noting the diaphragm's ability to recover.
  Assess the residual contraction of the diaphragm after mechanical ventilation to understand its recovery ability.
Diaphragmatic Displacement Velocity and Maximum Displacement | At each flow setting change: Measure the diaphragm's displacement velocity and maximum displacement at each HFNC flow rate adjustment.
  Displacement Velocity: The speed at which the diaphragm moves during each breath cycle.
  Maximum Displacement: The maximum distance the diaphragm moves during inhalation and exhalation.
Diaphragmatic ultrasound parameters (maximum displacement, thickening fraction, etc.) | At baseline (upon enrollment), 1 hour / 6 hours / 24 hours after the intervention, and daily morning assessments until extubation or day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Huiqing Ge, Study Chair — Sir Run Run Shaw Hospital
Locations (2):
- China (2):
  - Sir Run Run shaw Hospital Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goutman SA, Hamilton JD, Swihart B, Foerster B, Feldman EL, Rubin JM. Speckle tracking as a method to measure hemidiaphragm excursion. Muscle Nerve. 2017 Jan;55(1):125-127. doi: 10.1002/mus.25380. Epub 2016 Aug 22. PMID 27533320
- [Background] Santana PV, Cardenas LZ, Albuquerque ALP. Diaphragm Ultrasound in Critically Ill Patients on Mechanical Ventilation-Evolving Concepts. Diagnostics (Basel). 2023 Mar 15;13(6):1116. doi: 10.3390/diagnostics13061116. PMID 36980423
- [Background] Li R, Zhou Y, Chen W, Lyu L, Qiu G, Pan C, Tang Y. Speckle tracking ultrasound as a new tool to predict the weaning outcome of mechanical ventilation patients: a prospective observational study. Front Med (Lausanne). 2024 Dec 6;11:1449938. doi: 10.3389/fmed.2024.1449938. eCollection 2024. PMID 39712177
- [Background] Ye X, Liu Z, Ma Y, Song Y, Hu L, Luo J, Xiao H. A Novel Normalized Cross-Correlation Speckle-Tracking Ultrasound Algorithm for the Evaluation of Diaphragm Deformation. Front Med (Lausanne). 2021 Mar 12;8:612933. doi: 10.3389/fmed.2021.612933. eCollection 2021. PMID 33777969
- [Background] van den Berg MJW, Heunks L, Doorduin J. Advances in achieving lung and diaphragm-protective ventilation. Curr Opin Crit Care. 2025 Feb 1;31(1):38-46. doi: 10.1097/MCC.0000000000001228. Epub 2024 Nov 14. PMID 39560149
- [Background] Watanabe S, Sekiguchi K, Suehiro H, Yoshikawa M, Noda Y, Kamiyama N, Matsumoto R. Decreased diaphragm moving distance measured by ultrasound speckle tracking reflects poor prognosis in amyotrophic lateral sclerosis. Clin Neurophysiol Pract. 2024 Oct 22;9:252-260. doi: 10.1016/j.cnp.2024.10.002. eCollection 2024. PMID 39534515
- [Background] Xu Q, Yang X, Qian Y, Hu C, Lu W, Cai S, Hu B, Li J. Comparison of assessment of diaphragm function using speckle tracking between patients with successful and failed weaning: a multicentre, observational, pilot study. BMC Pulm Med. 2022 Dec 1;22(1):459. doi: 10.1186/s12890-022-02260-z. PMID 36456940
- [Background] Goligher EC, Jonkman AH, Dianti J, Vaporidi K, Beitler JR, Patel BK, Yoshida T, Jaber S, Dres M, Mauri T, Bellani G, Demoule A, Brochard L, Heunks L. Clinical strategies for implementing lung and diaphragm-protective ventilation: avoiding insufficient and excessive effort. Intensive Care Med. 2020 Dec;46(12):2314-2326. doi: 10.1007/s00134-020-06288-9. Epub 2020 Nov 2. PMID 33140181
- See also: Related Info — https://ccforum.biomedcentral.com/articles/10.1186/s13054-022-03975-5